CLINICAL TRIAL: NCT04586686
Title: Combining Interventions of Fertility Preservation to Mitigate Fertility Loss After
Brief Title: Combining Interventions of Fertility Preservation to Mitigate Fertility Loss After Breast Cancer
Acronym: Coimbra
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Hopital Antoine Beclere (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019COIMBRA001
Record Dates: First submitted 2020-08-11; First posted 2020-10-14 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer Female
Keywords: Fertility Preservation; Reproductive Techniques, assisted; Ovulation Induction; Oocyte Retrieval; Cryopreservation; Ovary
MeSH Terms: conditions — Helping Behavior

STUDY DESIGN:
Intervention Model Description: All patients will undergo a laparoscopy for an ovarian biopsy (about 20% of the ovarian volume). The side of the ovarian biopsy will be randomized on the day of the laparoscopy either from the right side (group 1) or from the left side (group 2). All patients will then continue with a controlled ovarian stimulation, using corifollitropin alpha and follitropin beta in a GnRH antagonist protocol using ganirelix. The metaphase II oocyte yield will be evaluated between the biopsied versus non-biopsied ovary to proof a non-inferiority (assuming that a difference of 1 metaphase II oocyte yielded from the biopsied ovary compared to the non-biopsied ovary is not clinically relevant).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: right ovarian biopsy (Other): Patients in group 1 will undergo a laparoscopy for an ovarian biopsy from the right ovary. They will then continue with a controlled ovarian stimulation, using a GnRH antagonist protocol. This will be started with Corifollitropin alfa 0.15 mg in the evening. On day six the antagonist, Ganirelix, will be added in the morning. If needed stimulation can be continued after seven days using follitropin beta daily in the evening (dosage ranging from 200-300 IE depending on AMH levels). Agonist trigger Triptorelin 0.2 mg will be administered for ovulation induction. In case of LH levels <2 IU/L at the start of ovarian stimulation, a dual ovulation strategy will be adapted: Triptorelin 0.2mg and choriongonadotropin 2500 IU (or choriongonadotropin alfa 250 µg) will be given. A transvaginal oocyte retrieval will be planned 36 hours after triggering.
  Interventions: Procedure: Ovarian biopsy via laparoscopy; Procedure: Transvaginal oocyte retrieval
- Group 2: left ovarian biopsy (Other): Patients in group 2 will undergo a laparoscopy for an ovarian biopsy from the left ovary. They will then continue with a controlled ovarian stimulation, using a GnRH antagonist protocol. This will be started with Corifollitropin alfa 0.15 mg in the evening. On day six the antagonist, Ganirelix, will be added in the morning. If needed stimulation can be continued after seven days using follitropin beta daily in the evening (dosage ranging from 200-300 IE depending on AMH levels). Agonist trigger Triptorelin 0.2 mg will be administered for ovulation induction. In case of LH levels <2 IU/L at the start of ovarian stimulation, a dual ovulation strategy will be adapted: Triptorelin 0.2mg and choriongonadotropin 2500 IU (or choriongonadotropin alfa 250 µg) will be given. A transvaginal oocyte retrieval will be planned 36 hours after triggering.
  Interventions: Procedure: Ovarian biopsy via laparoscopy; Procedure: Transvaginal oocyte retrieval

INTERVENTIONS:
Procedure: Ovarian biopsy via laparoscopy — A laparoscopy will be performed to achieve an ovarian cortical biopsy of one of both ovaries. Approximately twenty % of the ovarian volume as initially measured on the baseline ultrasound at the first visit will be removed to be processed in the lab for cortex freezing. The laparoscopic procedure in order to take the ovarian cortex biopsy will be standardised as much as possible. The technique developed by ProFam will be followed and adapted if needed by the surgeon's discretion. A three to four port laparoscopy will be used. The ovarian cortex biopsy will be taken using a curved scissor. Bipolar or unipolar cauterisation will be avoided as much as possible. If necessary for approximation or for hemostatic reasons, the ovarian edges can be stitched or Surgicel ® Absorbable Hemostat can be used.
Procedure: Transvaginal oocyte retrieval — After ovarian stimulation, a transvaginal oocyte retrieval will be performed either under local or general anaesthetics (patient's choice). The oocyte yield between the biopsied and non-biopsied ovary will be evaluated.

SUMMARY:
This clinical prospective randomised controlled trial will evaluate the impact of an ovarian biopsy on the oocyte yield after controlled ovarian stimulation before chemotherapy in view of breast cancer. The purpose of this trial is to learn about the possibility to combine these two fertility preservation procedures without decreasing the number of oocytes collected after an ovarian stimulation.

DETAILED DESCRIPTION:
All patients will undergo a biopsy of the ovarian cortex via laparoscopy, after patient eligibility has been established and patient consent has been obtained. The side of the ovarian biopsy will be randomized on the day of the laparoscopy either from the right side (group 1) or from the left side (group 2). The ovarian tissue will be cryopreserved. A small part will also be evaluated by the pathologist to screen for malignant contamination and follicle density. All patients will then continue with a controlled ovarian stimulation.

In both groups, a first blood analysis with hormonal assessment (E2, P, LH, FSH, hCG and AMH) will be performed at first visit, independent of their cycle. At that time a transvaginal ultrasound (frequency ≥ 7 MHz) will be done as well to assess the antral follicle count and the ovarian volume. The antral follicle count will be assessed using real-time 2D-US evaluation, the standard use in clinical practice. The ovarian volume will be measured using the prolate ellipsoid formula (volume = length x width x height x 0.523). If a dominant follicle is noted, choriongonadotropin (Pregnyl ® 5000 IU), choriongonadotropin Alfa (Ovitrelle ® 250 µg) or triptorelin (Gonapeptyl ® or Decapeptyl ® 0.2 mg) will be given to the patient to trigger ovulation. Thereafter, the controlled ovarian stimulation can be initiated in the luteal phase.

The size of the ovarian cortex biopsy will be calculated as 20% of the ovarian volume measured at the initial ultrasound. Immediately after the ovarian biopsy, the objective measurements of the biopsy will be noted in weight (gram) and volume (length x width x height mm³) because the biopsy fragment can be considered a rectangular box. A correction factor will be used afterwards in the statistical analysis if the volume of the ovarian biopsy is not equal to 20%.

The laparoscopic procedure by which the ovarian cortex biopsy will be performed, will be standardised: The technique developed by ProFam will be used and adapted if needed at the surgeon's discretion. A three to four-port laparoscopy will be used. The ovarian cortex biopsy will be performed using a curved scissor. Bipolar or unipolar cauterisation will be avoided as much as possible. If necessary for approximation or for hemostatic reasons, the ovarian edges can be stitched or Surgicel® Absorbable Hemostat can be used.

During the course of the study, there will be a number of blood analyses and ultrasounds, to evaluate follicular growth. This will be arranged at specific time points starting from day 6 of the stimulation and will be performed every other day, until the day of trigger. If necessary and based on clinician's decision, a supplementary blood analysis and/or ultrasound can be scheduled. At the follow-up ultrasounds the follicular growth will be noted for each ovary separately to assess difference in reaction and/or growth after the ovarian biopsy.

The controlled ovarian stimulation will start the day of the laparoscopy. It can start either in basal circumstances, or in the early follicular or luteal phase. A fixed GnRH antagonist protocol will be used. Ovarian stimulation will be started with Corifollitropin alfa 0.15 mg (Elonva®). On day six the antagonist, Ganirelix (Orgalutran®), will be added to prevent a premature LH surge. If needed ovarian stimulation can be continued after seven days using follitropin beta (Puregon®). The dosage of Puregon® is dependent on the AMH level at the first visit. Patients with AMH > 2 µg/L, will be started with 200-225 IE Puregon® daily. If the initial AMH level is <2 µg/L, patients will receive 225-300 IE Puregon® daily. Elonva ® and Puregon ® will be administered in the evening, whereas Orgalutran ® will be injected in the morning. Agonist trigger Triptorelin 0.2 mg (Gonapeptyl®) will be ministered as soon as at least three follicles reach a mean diameter of 18 mm or wider, with intermediary follicles 14 mm or wider. In case of LH levels <2 IU/L at the start of ovarian stimulation, a dual ovulation strategy will be adapted: Triptorelin 0.2mg and hCG 2500 IU (or ovitrelle 250 µg) will be given. Oocyte retrieval will be planned 36 hours after triggering. This will be performed as a transvaginal oocyte pick-up. Oocyte vitrification will be carried out after denudation and assessment of maturity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 35 years
* BMI ≥ 18 and ≤ 35 kg/m²
* Diagnosis of breast cancer
* Presence of 2 ovaries
* Signed informed consent form
* Medically fit for general anesthesia (ASA score 1-3)
* Permission of oncology team (with agreement to postpone chemo/radiotherapy for at least 2 weeks)
* Random start controlled ovarian stimulation
* AFC minimum (ie antral follicles measuring between 2-9 mm): 8 antral follicles

Exclusion Criteria:

* Age <18 or >35 years
* BMI <18 or >35 kg/m²
* Difference in AFC between the ovaries of more than 7 antral follicles
* Diagnosis of PCOS
* Previous radiotherapy and/or chemotherapy (neo-adjuvant chemotherapy included)
* Endometriose rAFS 3-4
* Allergy or reaction to the use of Elonva®, Puregon®, Orgalutran®, Pregnyl® Gonapeptyl®, Decapeptyl® or letrozole in the past

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mature oocyte yield from biopsied versus non-biopsied ovary | Immediately after the procedure of the transvaginal oocyte retrieval
  Evaluation of metaphase II oocyte yield between biopsied and non-biopsied ovary

SECONDARY OUTCOMES:
Follicle Output Rate (FORT) | From ovarian stimulation until the day of oocyte retrieval (2-3 weeks, depending on patient's response)
  Evaluation of the proportion of follicles that were responsive to FSH and is calculated by dividing the number of preovulatory follicles (16-20 mm) × 100 by the antral follicle count (3-8 mm)
COC yield | During the procedure of the transvaginal oocyte retrieval
  Evaluation of cumulus oophorus complex yield between biopsied and non-biopsied ovary
Maturation Rate | Immediately after the procedure of the transvaginal oocyte retrieval
  Evaluation of proportion of metaphase II oocytes within the COC yield between biopsies and non-biopsied ovary

CONTACTS AND LOCATIONS:
Overall Officials: Michel De Vos, MD PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (2):
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Brussels
  - UZ Gent, Ghent

IPD SHARING:
Plan to Share IPD: Yes
As this is a multicenter study, we plan to share IPD between the study sites. An electronical case report form (eCRF) will be set up and completed in all sites. Data will be handled in accordance with the general data protection regulation (GDPR).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available over the course of the study until 6 months after ending this study. This will give us the time to analyse the data of the different sites.
Access Criteria: eCRF

REFERENCES:
- [Background] De Vos M, Smitz J, Woodruff TK. Fertility preservation in women with cancer. Lancet. 2014 Oct 4;384(9950):1302-10. doi: 10.1016/S0140-6736(14)60834-5. PMID 25283571
- [Background] Garcia-Velasco JA, Domingo J, Cobo A, Martinez M, Carmona L, Pellicer A. Five years' experience using oocyte vitrification to preserve fertility for medical and nonmedical indications. Fertil Steril. 2013 Jun;99(7):1994-9. doi: 10.1016/j.fertnstert.2013.02.004. Epub 2013 Mar 1. PMID 23465707
- [Background] Decanter C, Cloquet M, Dassonneville A, D'Orazio E, Mailliez A, Pigny P. Different patterns of ovarian recovery after cancer treatment suggest various individual ovarian susceptibilities to chemotherapy. Reprod Biomed Online. 2018 Jun;36(6):711-718. doi: 10.1016/j.rbmo.2018.02.004. Epub 2018 Mar 2. PMID 29523398
- [Background] Cobo A, Garcia-Velasco J, Domingo J, Pellicer A, Remohi J. Elective and Onco-fertility preservation: factors related to IVF outcomes. Hum Reprod. 2018 Dec 1;33(12):2222-2231. doi: 10.1093/humrep/dey321. PMID 30383235
- [Background] Practice Committee of the American Society for Reproductive Medicine. Electronic address: asrm@asrm.org. Fertility preservation in patients undergoing gonadotoxic therapy or gonadectomy: a committee opinion. Fertil Steril. 2019 Dec;112(6):1022-1033. doi: 10.1016/j.fertnstert.2019.09.013. PMID 31843073
- [Background] Donnez J, Dolmans MM. Fertility Preservation in Women. N Engl J Med. 2017 Oct 26;377(17):1657-1665. doi: 10.1056/NEJMra1614676. No abstract available. PMID 29069558
- [Background] Diaz-Garcia C, Domingo J, Garcia-Velasco JA, Herraiz S, Mirabet V, Iniesta I, Cobo A, Remohi J, Pellicer A. Oocyte vitrification versus ovarian cortex transplantation in fertility preservation for adult women undergoing gonadotoxic treatments: a prospective cohort study. Fertil Steril. 2018 Mar;109(3):478-485.e2. doi: 10.1016/j.fertnstert.2017.11.018. Epub 2018 Feb 7. PMID 29428307
- [Background] Deb S, Kannamannadiar J, Campbell BK, Clewes JS, Raine-Fenning NJ. The interovarian variation in three-dimensional ultrasound markers of ovarian reserve in women undergoing baseline investigation for subfertility. Fertil Steril. 2011 Feb;95(2):667-72. doi: 10.1016/j.fertnstert.2010.09.031. Epub 2010 Oct 25. PMID 20971465
- [Background] Ueland FR, Depriest PD, Desimone CP, Pavlik EJ, Lele SM, Kryscio RJ, van Nagell JR Jr. The accuracy of examination under anesthesia and transvaginal sonography in evaluating ovarian size. Gynecol Oncol. 2005 Nov;99(2):400-3. doi: 10.1016/j.ygyno.2005.06.030. Epub 2005 Aug 9. PMID 16084576
- [Background] Amorim CA, Leonel ECR, Afifi Y, Coomarasamy A, Fishel S. Cryostorage and retransplantation of ovarian tissue as an infertility treatment. Best Pract Res Clin Endocrinol Metab. 2019 Feb;33(1):89-102. doi: 10.1016/j.beem.2018.09.002. Epub 2018 Sep 13. PMID 31208678
- [Background] Rodgers RJ, Reid GD, Koch J, Deans R, Ledger WL, Friedlander M, Gilchrist RB, Walters KA, Abbott JA. The safety and efficacy of controlled ovarian hyperstimulation for fertility preservation in women with early breast cancer: a systematic review. Hum Reprod. 2017 May 1;32(5):1033-1045. doi: 10.1093/humrep/dex027. PMID 28333356
- [Result] Dolmans MM, Marotta ML, Pirard C, Donnez J, Donnez O. Ovarian tissue cryopreservation followed by controlled ovarian stimulation and pick-up of mature oocytes does not impair the number or quality of retrieved oocytes. J Ovarian Res. 2014 Aug 26;7:80. doi: 10.1186/s13048-014-0080-8. PMID 25296615